CLINICAL TRIAL: NCT04105010
Title: A Phase I/II, Open-Label, Multicentre Study to Investigate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of AZD4205 in Patients With Peripheral T Cell Lymphoma (PTCL)
Brief Title: Assessing An Oral Janus Kinase Inhibitor, AZD4205 as Monotherapy in Patients Who Have PTCL (JACKPOT8)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DZ2019J0005
Record Dates: First submitted 2019-09-18; First posted 2019-09-26 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Relapsed or Refractory Peripheral T Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- golidocitinib Group A (Experimental): Group A: Open label golidocitinib at dose A, once daily (Phase 1)
  Interventions: Drug: golidocitinib
- golidocitinib Group B (Experimental): Group B: Open label golidocitinib at dose B, once daily (Phase 1)
  Interventions: Drug: golidocitinib
- golidocitinib Group C (Experimental): Group C: Open label golidocitinib at a selected dose, once daily (Phase 1)
  Interventions: Drug: golidocitinib
- golidocitinib Group D (Experimental): Group D: Open label golidocitinib at the RP2D, once daily (Phase 2)
  Interventions: Drug: golidocitinib

INTERVENTIONS:
Drug: golidocitinib — golidocitinib will be administered orally as capsules. golidocitinib treatment will be continued until disease progression or intolerant adverse reactions
  Other Names: AZD4205

SUMMARY:
This is a multinational, non-randomized, open-label, Phase 1/2 clinical study to evaluate the safety, tolerability and anti-tumor efficacy of AZD4205 as monotherapy in patients with peripheral T cell lymphoma (PTCL), who have relapsed from or are refractory/intolerant to standard systemic treatment.

Phase 1 part:

Around 20~40 patients will be subsequently enrolled into 2 different dose ascending cohorts. Additional 10~20 patients may be enrolled to further explore a selected dose defined by dose escalation cohorts.

Phase 2 part:

After the recommended phase 2 dose (RP2D) is defined, a phase 2 single-arm open-label pivotal study will be conducted to assess anti-tumor efficacy and safety of AZD4205 at RP2D in patients with refractory or relapsed PTCL.

ELIGIBILITY:
Inclusion Criteria:

1. Obtained written informed consent
2. Patients must have histologically confirmed peripheral T-cell lymphoma according to the 2016 revision of the World Health Organization classiﬁcation of lymphoid neoplasms. Tumor samples are required for central pathology review to confirm the diagnosis.
3. Patients must have measurable disease according to the Lugano criteria.
4. Patients should be transplant-ineligible upon their entry into this study, and must have relapsed after or been refractory/intolerant to ≥ 1 (but not > 3) prior systemic therapy(ies) for PTCL.
5. Adequate bone marrow reserve and organ system functions.

Exclusion Criteria:

1. Any unsolved toxicity > Common Terminology Criteria for Adverse Events (CTCAE) grade 1 from previous anti-cancer therapy (except alopecia).
2. Active infections, active or latent tuberculosis.
3. Patients with severely decreased lung function.
4. History of heart failure or QT interval prolongation.
5. Central nervous system (CNS) or leptomeningeal lymphoma.
6. History of treatment with Janus kinase (JAK) or signal transducer and activator of transcription 3 (STAT3) inhibitor.
7. Patient has undergone an allogeneic stem cell transplant. Patient had autologous stem cell transplant within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, PhD, Principal Investigator — Samsung Medical Center
Locations (50):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - Winship Cancer Institute, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Epworth Hospital, East Melbourne
  - St Vincent's Hospital Melbourne, Fitzroy
  - Royal Hobart Hospital, Hobart
  - St George Hospital, Kogarah
  - Royal Perth Hospital, Perth
  - Westmead Hospital, Westmead
- China (31):
  - Beijing Cancer Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Sichuan University - West China Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - The Second Hospital of Dalian Medical University, Dalian
  - Guangdong Provincial People's Hospital, Guangzhou
  - NanFang Hospital of Southern Medical University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - The Second Hospital of Anhui Medical University, Hefei
  - Shandong Cancer Hospital, Jinan
  - The First Hospital of Lanzhou University, Lanzhou
  - Linyi Cancer Hospital, Linyi
  - Jiangxi Province Cancer Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Cancer Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Cancer Hospital, Zhengzhou
- South Korea (9):
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song Y, Malpica L, Cai Q, Zhao W, Zhou K, Wu J, Zhang H, Mehta-Shah N, Ding K, Liu Y, Li Z, Zhang L, Zheng M, Jin J, Yang H, Shuang Y, Yoon DH, Gao S, Li W, Zhai Z, Zou L, Xi Y, Koh Y, Li F, Prince M, Zhou H, Lin L, Liu H, Allen P, Roncolato F, Yang Z, Kim WS, Zhu J. Golidocitinib, a selective JAK1 tyrosine-kinase inhibitor, in patients with refractory or relapsed peripheral T-cell lymphoma (JACKPOT8 Part B): a single-arm, multinational, phase 2 study. Lancet Oncol. 2024 Jan;25(1):117-125. doi: 10.1016/S1470-2045(23)00589-2. Epub 2023 Dec 9. PMID 38092009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: DZ2019J0005 study includes 2 parts: Part A, the dose escalation and extension part (group A, B, C), and part B, dose expansion part (group D).
  51 and 120 participants were recruited in Part A and Part B respectively, based on physician referral at 31 sites in the U.S., Australia, China and South Korea. The first participant was enrolled on 10-Sep-2019 and the last participant was enrolled on 23-Aug-2023.
Pre-assignment Details: 171 enrolled participants met inclusion criteria and received study drug.
Groups:
- AZD4205 Group A: Group A: Open label AZD4205 at 150 mg, once daily (Phase 1)
  AZD4205: AZD4205 will be administered orally as capsules. AZD4205 treatment will be continued until disease progression or intolerant adverse reactions
- AZD4205 Group B: Group B: Open label AZD4205 at 250 mg, once daily (Phase 1)
  AZD4205: AZD4205 will be administered orally as capsules. AZD4205 treatment will be continued until disease progression or intolerant adverse reactions
- AZD4205 Group C: Group C: Open label AZD4205 at 150 mg, once daily (Phase 1)
  AZD4205: AZD4205 will be administered orally as capsules. AZD4205 treatment will be continued until disease progression or intolerant adverse reactions
- AZD4205 Group D: Group D: Open label AZD4205 at the 150 mg (RP2D), once daily (Phase 2)
  AZD4205: AZD4205 will be administered orally as capsules. AZD4205 treatment will be continued until disease progression or intolerant adverse reactions
Period: Overall Study
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Started | 28 | 16 | 7 | 120
Completed | 13 | 7 | 5 | 39
Not Completed | 15 | 9 | 2 | 81
Not completed — Death | 3 | 1 | 1 | 54
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 8 | 1 | 1 | 4
Not completed — Other reason | 4 | 7 | 0 | 19

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (all patients treated with at least one dose of AZD4205)
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D | Total
Number analyzed (Participants) | 28 | 16 | 7 | 120 | 171
Age, Continuous [Median (Full Range); unit: years] | 62.5 [33 to 78] | 61.5 [29 to 79] | 55.0 [39 to 74] | 58.0 [20 to 79] | 58.0 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 3 | 44 | 61
  Male | 17 | 13 | 4 | 76 | 110
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 28 | 16 | 7 | 100 | 151
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 4 | 4
  White | 0 | 0 | 0 | 14 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part B: CT-based Objective Response Rate (ORR) by Independent Review Committee (IRC)
Description: ORR is the percentage of patients with at least one visit response of Complete Response (CR) or Partial Response (PR) based on CT scans evaluated by IRC per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Evaluable for CT-based Response Set (all dosed and central pathology confirmed Peripheral T Cell Lymphoma (PTCL) patients with baseline measurable disease assessed by IRC using CT imaging)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- AZD4205 Group D: Group D: Open label AZD4205 at 150 mg (RP2D), once daily (Phase 2)
  AZD4205: AZD4205 will be administered orally as capsules. AZD4205 treatment will be continued until disease progression or intolerant adverse reactions
Arm/Group | AZD4205 Group D
Number analyzed (Participants) | 102
percentage of participants | 43.1 [33.4 to 53.3]
Statistical Analysis 1: Comparison: AZD4205 Group D; Test type: Superiority; p < 0.0001, Binomial test against a null

2. Secondary Outcome: Part A and Part B: Number of Participants With Adverse Events
Description: To evaluate the safety and tolerability of AZD4205 in patients with PTCL in terms of adverse events (AEs), such as number of participants with AEs
Time Frame: The first dose until 28 days after last dose, up to approximately 3 years
Measure: Count of Participants; unit: Participants
Groups:
- AZD4205 Group D: Group D: Open label AZD4205 at the RP2D, once daily (Phase 2)
  AZD4205: AZD4205 will be administered orally as capsules. AZD4205 treatment will be continued until disease progression or intolerant adverse reactions
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 28 | 16 | 7 | 120
Participants | 26 | 16 | 6 | 115

3. Secondary Outcome: Part B: Duration of Response (DoR) Assessed by IRC
Description: DoR is the time from the date of first documented response until the date of documented progression or death due to any cause. Documented response and progression are both identified based on CT scans evaluated by IRC per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Subset of CR or PR responders in Evaluable for CT-based Response Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD4205 Group D
Number analyzed (Participants) | 44
months | NA [16.6 to NA] — Not estimable due to insufficient number of participants with events

4. Secondary Outcome: Part B: Complete Response Rate (CRR) Assessed by IRC
Description: CRR is the percentage of patients with at least one visit response of CR based on CT scans evaluated by IRC per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Evaluable for CT-based Response Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZD4205 Group D
Number analyzed (Participants) | 102
percentage of participants | 21.6 [14.0 to 30.8]

5. Secondary Outcome: Part B: Progression Free Survival (PFS) Assessed by IRC
Description: PFS is the time from the date of first dosing until the date of objective disease progression or death (by any cause) regardless of whether the participant discontinues the study treatments. Progression is identified based on CT scans evaluated by IRC per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Evaluable for Survival Set (all dosed and central pathology confirmed PTCL patients)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD4205 Group D
Number analyzed (Participants) | 105
months | 5.5 [3.0 to 18.7]

6. Secondary Outcome: Part B: Time to Response (TTR) Assessed by IRC
Description: TTR is the time from the date of first dosing to the time of the initial response of PR or CR. Response is identified based on CT scans evaluated by IRC per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Subset of CR or PR responders in Evaluable for CT-based Response Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD4205 Group D
Number analyzed (Participants) | 44
months | 1.4 [1.4 to 1.5]

7. Secondary Outcome: Part A and Part B: ORR Assessed by Investigator
Description: ORR is the percentage of patients with at least one visit response of CR or PR based on CT and/or PET scans evaluated by investigator per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Part A: Evaluable for Response Set (All dosed patients with baseline measurable disease) Part B: Evaluable for CT-based Response Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 28 | 16 | 7 | 102
percentage of participants | 46.4 [27.5 to 66.1] | 37.5 [15.2 to 64.6] | 14.3 [0.4 to 57.9] | 38.2 [28.8 to 48.4]

8. Secondary Outcome: Part A and Part B: DoR Assessed by Investigator
Description: DoR is the time from the date of first documented response until the date of documented progression or death due to any cause. Documented response and progression are both identified based on CT and/or PET scans evaluated by investigator per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Part A: Subset of CR or PR responders in Evaluable for Response Set Part B: Subset of CR or PR responders in Evaluable for CT-based Response Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 13 | 6 | 1 | 39
months | 5.09 [2.04 to NA] — Not estimable due to insufficient number of participants with events | NA [2.07 to NA] — Not estimable due to insufficient number of participants with events | 3.19 [NA to NA] — Not estimable due to insufficient number of participants with events | NA [4.4 to NA] — Not estimable due to insufficient number of participants with events

9. Secondary Outcome: Part A and Part B: CRR Assessed by Investigator
Description: CRR is the percentage of patients with at least one visit response of CR based on CT and/or PET scans evaluated by investigator per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Part A: Evaluable for Response Set Part B: Evaluable for CT-based Response Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 28 | 16 | 7 | 102
percentage of participants | 28.6 [13.2 to 48.7] | 12.5 [1.6 to 38.3] | 14.3 [0.4 to 57.9] | 14.7 [8.5 to 23.1]

10. Secondary Outcome: Part A and Part B: PFS Assessed by Investigator
Description: PFS is the time from the date of first dosing until the date of objective disease progression or death (by any cause) regardless of whether the participant discontinues the study treatments. Progression is identified based on CT and/or PET scans evaluated by investigator per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Part A: Safety Analysis Set Part B: Evaluable for Survival Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 28 | 16 | 7 | 105
months | 3.29 [1.31 to 3.58] | 2.50 [1.41 to NA] — Not estimable due to insufficient number of participants with events | 3.32 [1.41 to 5.26] | 3.4 [1.7 to 5.6]

11. Secondary Outcome: Part B: TTR Assessed by Investigator
Description: TTR is the time from the date of first dosing to the time of the initial response of PR or CR. Response is identified based on CT scans evaluated by investigator per Lugano criteria.
Time Frame: Up to approximately 3 years
Population: Subset of CR or PR responders in Evaluable for CT-based Response Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD4205 Group D
Number analyzed (Participants) | 39
months | 1.4 [1.4 to 1.5]

12. Secondary Outcome: Part A and Part B: Maximum Plasma Concentration (Cmax) of AZD4205
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data. Calculated for the single dose.
Time Frame: Cycle 1 Day 1 (each cycle = 21 days): 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 24 hours postdose (for Group A, B and C); 0 (predose), 1, 2, 4, 6, 8, and 24 hours postdose (for Group D).
Population: PK population (all dosed patients with at least one reportable AZD4205 plasma concentrations and no important AEs or protocol deviations that may impact PK) with Intensive PK sampling on Cycle 1, Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 27 | 16 | 7 | 38
ng/mL | 279.8 (29.2) | 512.0 (27.7) | 258.8 (36.9) | 229.2 (40.91)

13. Secondary Outcome: Part A and Part B: Area Under the Plasma Concentration-time Curve From Zero to the Last Measurable Concentration (AUC0-t) of AZD4205
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point, calculated by the linear up/log down rule.
Time Frame: Cycle 1, Day 1 (each cycle = 21 days): 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 24 hours postdose (for Group A, B and C); 0 (predose), 1, 2, 4, 6, 8, and 24 hours postdose (for Group D).
Population: PK population with Intensive PK sampling on Cycle 1, Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 27 | 16 | 7 | 38
h*ng/mL | 3592 (26.0) | 6755 (25.0) | 3276 (21.1) | 3271 (35.24)

14. Secondary Outcome: Part A and Part B: Cmax,ss, at Steady State of AZD4205
Description: Maximum observed plasma concentration (ng/mL) at steady state, obtained directly from the observed concentration versus time data. Calculated for the multiple doses.
Time Frame: Cycle 2 Day 1 (each cycle = 21 days): 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 24 hours postdose (for Group A, B and C); 0 (predose), 1, 2, 4, 6, 8, and 24 hours postdose (for Group D).
Population: PK population with Intensive PK sampling on Cycle 2, Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 20 | 7 | 6 | 23
ng/mL | 673.5 (28.9) | 1152 (30.6) | 665.9 (27.4) | 539.0 (35.92)

15. Secondary Outcome: Part A and Part B: AUCss, at Steady State of AZD4205
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point at steady state, calculated by the linear up/log down rule
Time Frame: as for outcome 14
Population: PK population with Intensive PK sampling on Cycle 2, Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
Number analyzed (Participants) | 20 | 7 | 6 | 23
h*ng/mL | 11978 (27.1) | 20991 (33.5) | 11822 (29.2) | 10000 (36.85)

ADVERSE EVENTS:
Time Frame: The first dose until 28 days after last dose, up to approximately 3 years
Arm/Group | AZD4205 Group A | AZD4205 Group B | AZD4205 Group C | AZD4205 Group D
All-Cause Mortality (participants affected / at risk) | 3/28 | 2/16 | 1/7 | 54/120
Serious Adverse Events (participants affected / at risk) | 12/28 | 9/16 | 1/7 | 44/120
Other Adverse Events (participants affected / at risk) | 26/28 | 16/16 | 6/7 | 114/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4205 Group A (N=28) | AZD4205 Group B (N=16) | AZD4205 Group C (N=7) | AZD4205 Group D (N=120)
Pneumonia (Infections and infestations) | 2 | 3 | 0 | 6
herpes zoster (Infections and infestations) | 0 | 0 | 0 | 4
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 | 0 | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 1 | 0 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Necrotising retinitis (Eye disorders) | 0 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 0 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypersplenism (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
death (General disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4205 Group A (N=28) | AZD4205 Group B (N=16) | AZD4205 Group C (N=7) | AZD4205 Group D (N=120)
Platelet count decreased (Investigations) | 9 | 7 | 0 | 71
Neutrophil count decreased (Investigations) | 6 | 7 | 1 | 62
White blood cell count decreased (Investigations) | 6 | 4 | 1 | 62
Lymphocyte count decreased (Investigations) | 5 | 0 | 0 | 36
Aspartate aminotransferase increased (Investigations) | 6 | 4 | 1 | 33
Alanine aminotransferase increased (Investigations) | 6 | 3 | 1 | 28
Blood lactate dehydrogenase increased (Investigations) | 1 | 3 | 0 | 25
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 20
Blood fibrinogen decreased (Investigations) | 1 | 2 | 2 | 17
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 16
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 12
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 10
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 8
Blood bilirubin increased (Investigations) | 2 | 1 | 1 | 7
Weight increased (Investigations) | 2 | 1 | 0 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 20
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 18
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 14
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 3 | 0 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2 | 0 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 7
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 2 | 51
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 7
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 15
Herpes zoster (Infections and infestations) | 1 | 2 | 0 | 13
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 13
Constipation (Gastrointestinal disorders) | 6 | 0 | 0 | 9
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 9
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 7
Nausea (Gastrointestinal disorders) | 5 | 1 | 0 | 7
Pyrexia (General disorders) | 9 | 6 | 1 | 24
Fatigue (General disorders) | 1 | 3 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 10
protein urine present (Investigations) | 0 | 2 | 0 | 5
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0 | 4
Blood chloride decreased (Investigations) | 0 | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 1
Epstein-Barr virus test positive (Investigations) | 0 | 1 | 0 | 1
Lung diffusion test decreased (Investigations) | 0 | 1 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 1 | 0 | 0
Prothrombin time shortened (Investigations) | 0 | 2 | 0 | 0
Pulmonary function test decreased (Investigations) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 1 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 2 | 3 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 0 | 10
Urinary tract infection (Infections and infestations) | 3 | 1 | 1 | 8
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 4
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2
Skin infection (Infections and infestations) | 0 | 1 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 1
Urethritis (Infections and infestations) | 2 | 0 | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 5
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 1
Facial pain (General disorders) | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 6
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 3 | 2 | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 3
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0 | 5
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 4
weight decreased (Investigations) | 0 | 1 | 0 | 6
urinary occult blood positive (Investigations) | 1 | 2 | 0 | 3
neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 9
white blood cell count increased (Investigations) | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT04105010/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT04105010/SAP_001.pdf